CLINICAL TRIAL: NCT04141904
Title: The Effects of the Anti-inflammatory Drug, Tofacitinib on Emotional and Reward Processing in Patients With Treatment-resistant Depression and Elevated High-sensitivity C-reactive Protein
Brief Title: Tofacitinib in Depression (TIDE)
Acronym: TIDE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Philip John Cowen, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19/SC/0136
Record Dates: First submitted 2019-10-14; First posted 2019-10-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Depression; Inflammation
Keywords: Depression
MeSH Terms: conditions — Depression; Inflammation | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups (tofacitinib or placebo) and take the assigned medication for 7-10 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tofacitinib (Experimental): Tofacitinib 5mg capsule twice a day for 7-10 days
  Interventions: Drug: Tofacitinib 5 MG [Xeljanz]
- Placebo (Placebo Comparator): Placebo capsule twice a day for 7-10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tofacitinib 5 MG [Xeljanz] — Tofacitinib 5mg capsules twice a day for 7-10 days
  Arms: Tofacitinib
Other: Placebo — Placebo capsules twice a day for 7-10 days
  Arms: Placebo

SUMMARY:
This study will test whether 7-10 day administration of the anti-inflammatory drug, tofacitinib, has positive effects on people experiencing treatment-resistant depression compared to placebo.

DETAILED DESCRIPTION:
This study uses a double-blind, placebo-controlled, randomised between groups design to test the hypothesis that, compared to placebo, 7-10 days' administration of tofacitinib 5mg twice daily has positive effects on emotional and reward processing in patients with treatment-resistant depression (TRD) and elevated C-reactive protein (hs-CRP; a marker of inflammation). Patients will have been diagnosed with Major Depressive Disorder using the Structured Clinical Interview for DSM-5 and will have shown non-response to at least 2 adequate antidepressant trials.They will also have a plasma hs-CRP of 1mg/L or greater. During the study patients will continue their antidepressant treatment. Participants will be randomised to receive 7-10 days treatment with either tofacitinib 5 mg twice daily or a matched placebo. This study includes three visits in total: a screening visit; research visit 1 (includes cognitive tests) and research visit 2 (to include an MRI scan as well as cognitive tests).

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Aged 18-65 years;
* Willing and able to give informed consent for participation in the study;
* Sufficiently fluent English to understand and complete the tasks;
* Registered with a GP and consents to GP being informed of participation in the study;
* Participants need to meet a number of concurrent clinical criteria:
* Current criteria for Major Depressive Disorder [as determined by the Structured Clinical interview for DSM-5 (SCID-5)];
* Inadequate response to at least two adequate courses of antidepressant therapy each given at a therapeutic dose for at least four weeks;
* Baseline elevated inflammation [as determined by high-sensitivity C-reactive protein (hs-CRP) of 1mg/L or greater [~70% of patients expected to be above (estimated from Chamberlain-2018)];
* Participants engaging in sex with a risk of pregnancy must agree to use a highly effective method of contraception from Screening Visit until 30 days after receiving the study medication treatment. Acceptable methods of contraception include:
* Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal;
* Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable or implantable;
* Intrauterine device (IUD);
* Intrauterine hormone-releasing system (IUS);
* Bilateral tubal occlusion;
* Vasectomy (or vasectomised partner);
* Condoms +/- spermicides;
* Sexual abstinence. [Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), and spermicides only are not acceptable methods of contraception.]
* Male participants must not donate sperm

Exclusion Criteria:

* History of /or current DSM-5 bipolar disorder or schizophrenia.
* Current DSM-5 eating disorder.
* Participants who fulfil current criteria for other comorbid disorders may still be entered into the study, if, in the opinion of the Investigator, the psychiatric diagnosis will not compromise safety or affect data quality;
* Participants currently taking strong cytochrome P450 (CYPs) 3A4 inhibitors (e.g. fluvoxamine)
* Electroconvulsive therapy for the treatment of the current episode of depression;
* Clinically significant abnormal values for full blood count, urea and electrolytes, liver function tests, blood pressure, or ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures;
* Participants who are positive for blood-borne viruses (HIV/HepB/HepC);
* Participants who are positive to tuberculosis' screening test (T-SPOT.TB +);
* Participants receiving or planning to receive a live vaccine within 4 weeks of study treatment; if the patient is due an influenza vaccine, this should be rescheduled to 2 weeks after the study.
* History of significant alcohol/substance misuse or dependence over the past 6 months;
* History of, or current medical conditions that in the opinion of the Investigator may interfere with the safety of the participant or the scientific integrity of the study, including recurrent infections (e.g. sinusitis, genital herpes simplex, or herpes zoster), malignancies (except for successfully treated non-melanoma skin cancer or localised carcinoma in situ of the cervix), severe neurological problems (e.g. Parkinson's disease; blackouts requiring hospitalization, epilepsy/seizures, stroke, other brain injury), severe cardiovascular disorder (e.g. moderate-severe congestive heart failure, cerebrovascular accident, myocardial infarction, coronary stenting, uncontrolled hypertension systolic >160 mmHg or diastolic >100 mmHg, unprovoked deep vein thrombosis or pulmonary embolism), severe haematological disorder (e.g. total white blood cell count <3,000/μL, absolute neutrophil count <1,500/μL, platelet count <100,000/μL, absolute lymphocyte count <800/μL, hemoglobin <10 g/dL), severe hepatic disease (e.g. serum alanine transaminase (ALT) >2 × upper limit of normal), significant renal disease (e.g. estimated glomerular filtration rate (GFR) by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula > 40 mL/min/1.73m2), severe gastro-intestinal problems (e.g. diverticulitis, previous perforation or high risk of perforation, conditions that could interfere with drug absorption including but not limited to short bowel syndrome); previous organ transplant;
* Clinically significant risk of suicide;
* Current pregnancy (as determined by urine pregnancy test taken during the Screening Visit and the Research Visit One), breastfeeding, or planning a pregnancy during the course of the study;
* Participants with Body Mass Index (BMI - kg/m2) outside the 18-36 range at Screening Visit;
* Participants with severe claustrophobia;
* Participants with ferromagnetic objects in their bodies (e.g. metal implants, vessel clips, shrapnel injuries) or with implanted devices which may be damaged by the magnet (e.g. heart pacemakers);
* Previous participation in a study using the same, or similar, emotional or reward processing tasks;
* Previous participation in a psychological or medical study involving the use of medication within the last 3 months;
* Participant received non-prescription medication, including supplements such as vitamins and herbal supplements within 48 hours prior to the Research Visit One (apart from paracetamol). Participants who have taken non-prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety;
* Participant with a known hypersensitivity to tofacitinib;
* Participant with planned medical treatment within the study period that might interfere with the study procedures;
* Participant who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
The effects of tofacitinib on emotional processing using the Facial Expression Recognition Task (FERT) | Day 7-10 of drug/placebo administration
  Accuracy and reaction times on computer-based tasks of emotional processing using facial expressions of basic emotions (happiness, fear, anger, disgust, sadness, surprise) are displayed on the screen and participants are asked to correctly classify them. Each emotion is presented at different intensity levels. Responses are made via a button-press and accuracy and reaction time are recorded

SECONDARY OUTCOMES:
The effects of tofacitinib on Emotional Memory Task (EMEM) scores | Day 7-10 of drug/placebo administration
  Recall and recognition of affective words displayed earlier in the testing session is tested
Emotional categorization using the Emotional categorization task (ECAT) | Day 7-10 of drug/placebo administration
  Disagreeable or agreeable personality descriptions are presented and participants are asked to indicate whether they would like or dislike to be described as each of these characteristics. Responses are made via a button-press.
Emotional recall task (EREC) | Day 7-10 of drug/placebo administration
  Participants are asked to write down as many of the words as they can remember from the previous task. Responses are made via pencil and paper.
Brain neural activity | Day 7-10 of drug/placebo administration
  BOLD fMRI at resting state and during the performance of an emotional (i.e. covert facial expression processing) and a reward (i.e. adapted probabilistic instrumental learning) processing tasks.
Faces dot probe task (FDOT) | Day 7-10 of drug/placebo administration
  Participants carry out computer-based tasks and attentional vigilance to happy or fearful faces is recorded from participants' response latency to indicate the alignment of a dot probe appearing in the place of one of the faces
Probabilistic Instrumental Learning Task (PILT) | Day 7-10 of drug/placebo administration
  Participants have to learn which shapes are associated with wins and losses and sensitivity to reward is measured.
Auditory Verbal Learning Task (AVLT) | Day 7-10 of drug/placebo administration
  Accuracy of recall on the auditory verbal learning task
The effects of tofacitinib on cerebral perfusion | Day 7-10 of drug/placebo administration
  Arterial spin labelling at rest to measure cerebral perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cowen, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided